CLINICAL TRIAL: NCT06586346
Title: Frequency, Predictors and Outcome of Sepsis Induced Coagulopathy in Critical Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira ahmed mohamed samony, Principal investigator, Assiut University
Other Study IDs: Sepsis induced coagulopathy
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In intensive care units , sepsis remains one of the common causes of mortality and morbidity . The average hospital length of stay for sepsis is twice as long as any other fatal condition . Furthermore, sepsis survivors are at an increased risk of death or a reduced health related quality of life even after discharge from the hospital . Sepsis induces multiple and complex derangements in many systems including the coagulation cascade. The vast majority of septic patients present with hemostatic abnormalities ranging from subclinical coagulopathy to fulminant disseminated intravascular coagulation . During the initial stages of infection coagulation operates as a natural defense mechanism attempting to confine the responsible pathogen and prevent its spread into systematic circulation. However in advanced and severe infections as in sepsis, mass inflammatory cytokine production and release into the circulation lead to significantly deranged hemostatic balance . The coagulation process is activated while anticoagulant mechanisms including fibrinolysis and anticoagulant factors are suppressed. Consequently septic patients are prone to a prothrombotic state through four main mechanisms extrinsic pathway activation, cytokine induced coagulation amplification, anticoagulant pathways suppression, and fibrinolysis impairment .

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening syndrome associated with physiological, pathological and biological abnormalities caused by a dysregulated host response to infections . Globally, there are ∼48.9 million sepsis cases, leading to 11 million deaths annually .

In intensive care units , sepsis remains one of the common causes of mortality and morbidity . The average hospital length of stay for sepsis is twice as long as any other fatal condition and the in-hospital mortality remains as high as 20% . Furthermore, sepsis survivors are at an increased risk of death or a reduced health-related quality of life even after discharge from the hospital .

Sepsis induces multiple and complex derangements in many systems, including the coagulation cascade. The vast majority of septic patients present with hemostatic abnormalities, ranging from subclinical coagulopathy to fulminant disseminated intravascular coagulation (DIC) . During the initial stages of infection, coagulation operates as a natural defense mechanism, attempting to confine the responsible pathogen and prevent its spread into systematic circulation. However, in advanced and severe infections, as in sepsis, mass inflammatory cytokine production and release into the circulation lead to significantly deranged hemostatic balance . The coagulation process is activated, while anticoagulant mechanisms, including fibrinolysis and anticoagulant factors, are suppressed. Consequently, septic patients are prone to a prothrombotic state through 4 main mechanisms: extrinsic pathway activation, cytokine-induced coagulation amplification, anticoagulant pathways suppression, and fibrinolysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of ago or older who will be admitted to critical care unit with sepsis during period between october 2024 and october 2026.

Exclusion Criteria:

* patients under tge age of 18patients with end organ diseases
* pregnant woman
* patient with coagulation disorder
* patient using anticoagulant drugs

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with 18 years of ago or older who will be admitted to critical care unit with sepsis during period between october 2024 and october 2026 ,they will divided into two groups according to development of sepsis induced coagulopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assess frequency and severity of sepsis induced coagulopathy in critical care unit | 10/9/2024 - 1/10/2026
  Assess frequency and severity of sepsis induced coagulopathy in critical care unit

CONTACTS AND LOCATIONS:
Overall Officials: Dina Ali, Dr, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No